CLINICAL TRIAL: NCT02229279
Title: Evaluation of Teleconsulting on Rehabilitation After Hip and Knee Surgical Procedures
Acronym: SSRHAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLM-HAD
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: Surgical Procedures, Operative
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teleconsulting (Active Comparator): Teleconsulting
  Interventions: Device: Teleconsulting
- No Teleconsulting (No Intervention)

INTERVENTIONS:
Device: Teleconsulting
  Other Names: Telemedicine
  Arms: Teleconsulting

SUMMARY:
The objective of this study is to assess the medical and economic relevance of teleconsulting for Rehabilitation After Hip and Knee Surgical Procedures.

ELIGIBILITY:
Inclusion Criteria:

* Post hip or knee surgery
* Fulfilment of criteria for home rehabilitation (no need for hospital treatment post surgery)

Exclusion Criteria:

* Social isolation
* Life threatening condition
* No GSM network
* No DSL network

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Functional subscore of simplified WOMAC Scale | up to 30 days after start of rehabilitation

SECONDARY OUTCOMES:
Joint Paint measured with visual analogue scale | up to 30 days after start of rehabilitation
Patient satisfaction questionnaire | The last 1 day of the rehabilitation
Medical and paramedical staff satisfaction questionnaire | 6 months after enrollment of the first patient
Overall costs of treatment | 6 months after enrollment of the first patient
Number of hospitalizations and use of emergency units | Within 30 days after start of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Copin, MD, Principal Investigator — Fondation Santé Service, Pôle Rééducation - Handicap; Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique - Hôpitaux de Paris
Locations (1):
- Fondation Santé Service, Pôle Rééducation- Handicap, Puteaux, France

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Background] Tubach F, Baron G, Falissard B, Logeart I, Dougados M, Bellamy N, Ravaud P. Using patients' and rheumatologists' opinions to specify a short form of the WOMAC function subscale. Ann Rheum Dis. 2005 Jan;64(1):75-9. doi: 10.1136/ard.2003.019539. PMID 15608303
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] Baron G, Tubach F, Ravaud P, Logeart I, Dougados M. Validation of a short form of the Western Ontario and McMaster Universities Osteoarthritis Index function subscale in hip and knee osteoarthritis. Arthritis Rheum. 2007 May 15;57(4):633-8. doi: 10.1002/art.22685. PMID 17471534
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558